CLINICAL TRIAL: NCT01392222
Title: Treatment Decision-Making Among Patients Diagnosed With Papillary Microcarcinoma and Their Significant Others
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-108
Record Dates: First submitted 2011-06-29; First posted 2011-07-12 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Thyroid Cancer; Papillary Microcarcinoma
Keywords: focus group; 11-108
MeSH Terms: conditions — Thyroid Neoplasms; Papillary Thyroid Microcarcinoma | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (2):
- patients who have had surgery or have scheduled surgery: In this exploratory study we will conduct focus groups and individual interviews with two population segments according to the established methodology of Krueger and Casey [13] and Morgan [14]. We will conduct 4-6 focus groups, two to three within each population segment, to evaluate the process of decision-making to manage papillary microcarcinoma, factors that influenced decision-making, understanding of risk for recurrence and other negative outcomes due to thyroid cancer, information needed to make informed decisions, and what could influence thyroid cancer patients who have had surgery or have scheduled to have surgery to remove their papillary microcarcinomas to consider active surveillance. Individual interviews will be offered and conducted as needed for those patients who are unable to attend a focus group due to scheduling conflicts or other reasons.
  Interventions: Behavioral: Focus groups
- who chose to not have immediate surgery: In this exploratory study we will conduct focus groups with two population segments according to the established methodology of Krueger and Casey [13] and Morgan [14]. We will conduct 4-6 focus groups, two to three within each population segment, to evaluate the process of decision-making to manage papillary microcarcinoma, factors that influenced decision-making, understanding of risk for recurrence and other negative outcomes due to thyroid cancer, information needed to make informed decisions, and what could influence thyroid cancer patients who have had surgery or have scheduled to have surgery to remove their papillary microcarcinomas to consider active surveillance. Individual interviews will be offered and conducted as needed for those patients who are unable to attend a focus group due to scheduling conflicts or other reasons.
  Interventions: Behavioral: Focus groups

INTERVENTIONS:
Behavioral: Focus groups — The focus groups will cover the following issues
  * Perceptions of thyroid cancer and disease status
  * Sources of information used in papillary microcarcinoma treatment decision-making
  * Treatment decision-making processes and influential factors
  * Perceived barriers to active surveillance to treat papillary microcarcinoma (for the immediate surgery sub-sample)
  * Perceived facilitators to active surveillance to treat papillary microcarcinoma (for the non-immediate surgery sub-sample)
  * Views about how to improve acceptability of active surveillance as a disease management option
  Other Names: Each focus group will last between approximately 90-120 minutes and each; individual interview will last approximately 60 minutes. Notes will be taken; during each focus group and individual interviews. All focus groups and; individual interviews, will be audio-recorded with digital voice recorders,; and the recordings will be transcribed by a professional transcription service,; for later qualitative analysis. Individual interviews will be offered to those; patients who are unable to attend a focus group due to scheduling conflicts or other reasons.; Participants interested in taking part in the optional member check will be mailed a summary; document created by the research team. A surgery group summary document will be mailed to; surgery patients and an active surveillance summary document will be mailed to active surveillance; patients. Each summary document will include data, analytic categories, interpretations, and; conclusions reached by the analytic team.
  Groups: patients who have had surgery or have scheduled surgery
Behavioral: Focus groups — The focus groups will cover the following issues:
  * Perceptions of thyroid cancer and disease status
  * Sources of information used in papillary microcarcinoma treatment decision-making
  * Treatment decision-making processes and influential factors
  * Perceived barriers to active surveillance to treat papillary microcarcinoma (for the immediate surgery sub-sample)
  * Perceived facilitators to active surveillance to treat papillary microcarcinoma (for the non-immediate surgery sub-sample)
  * Views about how to improve acceptability of active surveillance as a disease management option
  Other Names: Each focus group will last between approximately 90-120 minutes and each individual interview will; last approximately 60 minutes. All focus groups and individual interviews, will be audio-recorded; with digital voice recorders. Notes will be taken during each focus group and each individual interview; the recordings will be transcribed by, a professional transcription service,; for later qualitative analysis. Individual interviews will be offered to those; patients who are unable to attend a focus group due to; scheduling conflicts or other reasons.; Participants interested in taking part in the optional member check will be mailed a summary; document created by the research team. A surgery group summary document will be mailed to; surgery patients and an active surveillance summary document will be mailed to active surveillance; patients. Each summary document will include data, analytic categories, interpretations, and; conclusions reached by the analytic team.
  Groups: who chose to not have immediate surgery

SUMMARY:
The purpose of this study is to understand more about why some patients choose to have surgery to treat their papillary microcarcinoma (PMC) and others choose to have their papillary microcarcinoma (PMC) regularly watched by their doctor to see if and when they may need surgery (referred to as "active surveillance"). The investigators also hope learn more about what patients and their family members worry about or feel they will gain from surgery or active surveillance.

ELIGIBILITY:
Inclusion Criteria:

Thyroid cancer patient eligibility will include:

* Thyroid cancer patients who have been diagnosed with papillary microcarcinoma (or subcentimeter thyroid lesions with fine needle aspiration biopsy suspicious for papillary or follicular thyroid cancer) within the prior 6-12 months as per EMR path report and clinician assessment;
* Presented with the option of treating their papillary microcarcinomas with either surgery or active surveillance as per treating physician;
* English-fluent;
* 18 years of age or older;

Patient-designated significant other eligibility will include:

* Nomination by patient as individual who assisted patient in decision-making regarding how to treat thyroid papillary microcarcinoma;
* English-fluent;
* 18 years of age or older;

Exclusion Criteria:

Thyroid cancer patient exclusion criteria will include:

* Thyroid cancer patients with known loco-regional or distant metastases prior to initial surgical intervention as per path report.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants will be recruited from Dr. Mike Tuttle's clinic.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
To explore patients' and families' perceived risks and benefits of active surveillance and surgery within the context of papillary microcarcinoma. | 5 years
  We'll conduct focus groups & individual interviews with 2 population segments established by the method of Krueger & Casey & Morgan. The population segments will be thyroid cancer patients who have had surg or have scheduled surg, & any pt-designated significant others who assisted pts with tx decision-making & thyroid cancer pts who chose to not have immediate surg, whether they are either postponing their tx decision until a later date, or have committed to active surveillance rather than surg, & any pt-designated significant others who assisted these patients with tx decision-making.

SECONDARY OUTCOMES:
To examine the factors in patients' and families' decision making about the treatment of papillary microcarcinoma. | 5 years
  We'll conduct focus groups & individual interviews with 2 population segments established by the method of Krueger & Casey & Morgan. The population segments will be thyroid cancer pts who have had surg or have scheduled surg, & any pt-designated significant others who assisted patients with tx decision-making & thyroid cancer pts who chose to not have immediate surg, whether they are either postponing their tx decision until a later date, or have committed to active surveillance rather than surg, & any patient-designated significant others who assisted these pts with tx decision-making.

CONTACTS AND LOCATIONS:
Overall Officials: Smita Banerjee, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm